CLINICAL TRIAL: NCT04841499
Title: Effects of a Seven-day BASIS™ Supplementation on Menopausal Syndromes and Measurements of the Urinary Vitamin B3 and Estradiol Levels in Pre-, Peri- and Post-menopause
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of South Alabama (Other)
Collaborators: Elysium Health, Inc. (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: USAH-EH301
Record Dates: First submitted 2021-04-07; First posted 2021-04-12 (Actual); Last update posted 2021-11-18 (Actual); Status verified 2021-11

CONDITIONS: Menopause
Keywords: pre menopause, peri menopause, post menopause, menopause, hot flashes, declining estradiol leves
MeSH Terms: conditions — Hot Flashes | interventions — Pterocarpus marsupium

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment Arm (Experimental): 7 days of BASIS™ orally
  Interventions: Drug: BASIS™ (Crystalline Nicotinamide Riboside 250mg and Pterostilbene 50mg)

INTERVENTIONS:
Drug: BASIS™ (Crystalline Nicotinamide Riboside 250mg and Pterostilbene 50mg) — take 2 capsules orally each day for 7 days

SUMMARY:
The purpose of this study is to determine whether a short supplementation (7days) with BASIS™ increases the natural production of estradiol, measured in urinary waste. The overall objective is to determine whether through increased estradiol levels, the undesirable menopausal effects, assessed via questionnaires, are mitigated by a short-term supplementation with BASIS™

DETAILED DESCRIPTION:
Protocol Outline

Protocol Title: Effects of a seven-day BASIS™ supplementation on menopausal syndromes and measurements of the urinary vitamin B3 and estradiol levels in pre-, peri- and post-menopause.

I. Abstract

Context:

Nicotinamide adenine dinucleotide (NAD) is a derivative of vitamin B3 necessary to the production of key hormonal regulators like estradiol. As we age, both NAD levels and estradiol levels are reduced. Reduced estradiol levels have been associated with menopausal syndromes. BASIS™ recent clinical outcomes have shown that this NAD precursor (BASIS™) boosts declining NAD levels. In an n=1 study, repeated over 3 years, a short intake (<1week at 125mg/day) of over-the-counter nicotinamide riboside, one of the two active ingredients of BASIS™, by a peri-menopausal 50-year-old female, resulted in the blunting of the undesirable menopausal effects such as poor sleep and hot flashes. The other component of BASIS™ is pterostilbene, a phytoestrogen, derivative of resveratrol. Phytoestrogens associate with the protection of estradiol levels and relief of menopausal syndrome in women using over-the-counter phytoestrogens. These outcomes and observations have prompted the proposed study. We wish to establish whether the observed beneficial effects of nicotinamide riboside and the reported beneficial effects of phytoestrogens on menopausal syndromes can work synergistically with a product like BASIS™ and are observed more broadly in peri- and menopausal women. Furthermore, we wish to establish whether remediation of symptoms can be attributed to a naturally occurring increase in estradiol levels following the repletion of NAD by BASIS™.

Objectives:

The first objective is to determine whether a short supplementation with BASIS™ increases the natural production of estradiol, measured in urinary waste. The second objective is to determine whether, through increased estradiol levels, the undesirable menopausal effects are mitigated by a short-term supplementation with BASIS™.

Study Design:

Women suffering from undesirable menopause-related discomfort will be entered in this study. Discomfort includes mood swings, hot flashes, bad sleep, and dry skin. The control cohort will be composed of women who are pre-menopausal. All women entering the study will be given a questionnaire before taking BASIS™ and once they have completed the 7-day supplementation. They will also be asked to provide a urine sample at the time of each survey. The urine samples will be analyzed for total estradiol content (estradiol, sulfate and glucoronate, and estriol; all metabolites of estradiol) and for total vitamin B3 content.

II. Background and Significance/Preliminary Studies Menopause signals the end of the natural reproductive potential and declining hormone levels for women; hormones such as estradiol. Typically, a well-orchestrated sequence of estrogen, progesterone, and testosterone production occurs each month with ovulation, but as we age, sex hormone levels start to fluctuate and eventually decline significantly. This can last for upwards of 10 years prior to the last menstrual cycle (peri-menopause).

Our brain, muscle, liver, skin, and fat cells all have hormone receptors, thus as changes occur, they affect organ function on a cellular level. The climacteric syndrome is characterized by several symptoms: hot flashes are the most common and reported by about 70% of peri- post-menopausal women. Sleep disorders particularly decreased sleep quality, and irritability are also commonly reported. Common biological mechanisms may explain in part the relationship between hot flushes, sleep disorders, and irritability. For example, withdrawal of hormones causes a change in the serotonin levels. The serotonergic system is implicated in sleep, mood, and hot flashes. Tryptophan, an essential amino acid, is the precursor for serotonin synthesis. Critically, tryptophan is also a precursor to nicotinamide adenine dinucleotide, NAD[5]. NAD and its derivative NADPH are central cofactors to cellular metabolism and cellular signaling with critical roles in aging. They are also co-substrates in many biosynthetic pathways, including of estrogen-derived hormones such as estradiol. Increased oxidative stress and declining NAD levels would affect the biosynthetic pathways leading to estradiol[6]. Critically, estradiol levels steadily decrease over the course of peri and post-menopause; a process which has been correlated to the occurrence and intensity of menopausal symptoms (https://www.menopause.org/for-women/menopauseflashes/menopause-symptoms-and-treatments/the-experts-do-agree-about-hormone-therapy).

Recent investigations in the field of NAD and NADP have unveiled a range of biosynthetic, orally available precursors (nicotinamide riboside and nicotinamide mononucleotide), which are able to boost NAD levels systemically[7]. This has led to a vast number of clinical trials to investigate whether and if so by how much these precursors could boost circulating NAD and alleviate age-associated disorders, such a metabolic dysfunction, obesity and cellular aging. It has been suggested that oxidative stress, which increased NAD levels appears to remediate, may also play a role in sleep disorders. While the outcomes remain inconclusive in terms of clinical impact, these NAD precursors were shown to be safe and well-tolerated by numerous types of participants at dosages as high as 1gram/day. One of these trials included BASIS™. In addition to nicotinamide riboside, BASIS™ also includes pterostilbene in its formulation. Critically, resveratrol and pterostilbene have a similar chemical structure to the diethylstilbestrol and 17-beta estradiol and act as phytoestrogens, protectors of estradiol levels. Furthermore, estrogen-like entities, phytoestrogen are thought to enhance NAD function in cellular metabolism[8].

We hypothesize that as we age, a reduction in NAD levels and a shift in redox balance leading and causing oxidative stress could correlate to a decrease in the production of estradiol. This causation could be direct, by simply reducing the activity of the NAD(P) dependent enzymes involved in the synthesis of estradiol and its precursors or indirect by NAD-dependent protein post-translational modulation of gene expression pathways that impact estradiol biosynthesis and function. A nutraceutical approach that combines increased levels of NAD(P) to phytoestrogens like pterostilbene may be useful to preventive or at least moderate the intensity of the menopausal syndromes controlled by reduced estradiol levels.

III. Study Aims

This is a pilot study that seeks to enroll up to 40 female individuals over 35 years of age. The purpose of this study is to determine whether a short supplementation (7days) with BASIS™ increases the natural production of estradiol, measured in urinary waste. The overall objective is to determine whether through increased estradiol levels, the undesirable menopausal effects, assessed via questionnaires, are mitigated by a short-term supplementation with BASIS™

IV. Administrative Organization

The study will be administered at the MCI.

V. Study Design

1. Experimental design of the study: This is a single-arm study for which non-peri and non-menopausal women will act as a control cohort. We will seek for 25% of the recruited cohort to be within the control group.
2. Study population general description: Any healthy women older than 35years of age can partake in this study. However, individuals receiving hormone replacement therapy will be excluded from the study.
3. Sample size determination and power analyses: This is a pilot study to establish the proposed correlation between metabolites. Studies as small as 12 individuals have been conducted to establish pharmacological roles for nicotinamide riboside as well as for pterostilbene. Similar sample sizes have been employed to investigate the properties of exogenous estradiol on sleep quality and hot flashes[9].
4. The outcomes of the study are three folds:

   1. A correlation between levels of estradiol and bioavailability of circulating NAD boosted by nicotinamide riboside will be established.
   2. A correlation between NAD bioavailability and the occurrence and intensity of undesirable menopausal symptoms will be established.
   3. A correlation between the synergistic effect of NAD increase and pterostilbene on the occurrence and intensity of undesirable menopausal symptoms by naturally enhancing levels of estradiol will be established.

d. Study Assessments and Activities i. Following completion of the consent form, the participants will be asked to fill a pre-supplementation questionnaire. They then will be asked to provide a urinary sample after being given a urine sampling kit. Following this, the participant will be provided with a small jar of BASISTM (supplies≥7days). The participant will take 2 capsules of BASISTM once a day (total daily dose contains 250mg of nicotinamide riboside and 50mg of pterostilbene). After 7 days, the participants will be asked to provide a second urine in the urine sampling kit provided to them and fill in the same questionnaire.

ii. The questionnaire aims to evaluate the intensity and frequency of the most common menopause-associated undesirable symptoms.

iii. Provide a schedule of all study assessments and subject activities, including a tabular representation or timeline as applicable:

iv. Following completion of the consent form, the participants will be asked to fill in a pre-supplementation questionnaire. They then will be asked to provide a urinary sample after being given a urine sampling kit. Following this, the participant will be provided with a small jar of BASIS™ (supplies>7days). The participant will take 2 capsules of BASIS™ once a day (total daily dose contains 250 mg of nicotinamide riboside and 50 mg of pterostilbene). After 7 days, the participants will be asked to provide a second urine sample in the urine sampling kit provided to them and fill in the same questionnaire.

v. The questionnaire aims to evaluate the intensity and frequency of the most common menopause-associated undesirable symptoms.

vi. Provide a schedule of all study assessments and subject activities, including a tabular representation or timeline as applicable (visit chart in the full protocol)

VIII. Analysis Plan

This is a short-term metabolic study for which pharmacokinetics and pharmacodynamics outcomes are anticipated. There will be no intention-to-treat methodology in the analysis. There will be no sample stratification. The urine content of the NAD and estradiol catabolomes' measurements will be presented as mean of biological replicates and 95% confidence interval (CI) from all analyzed LC-MS measurements pooled from 2 technical replicates. For multiple comparisons, ANOVA followed by posthoc test, i.e., Bonferroni correction for LC-MS and Dunnett's or Tukey's for combination with questionnaire outcomes. Dependent t-tests and repeated measures ANOVA will be used to evaluate within sub-groups variability. Statistical analysis is performed using GraphPad PRISM 7.

DATA AND SAFETY MONITORING PLAN (DSMP):

INSTRUCTIONS FOR COMPLETION The purpose of this monitoring plan is to provide practical guidelines for clinical monitoring procedures and to ensure proper auditing of the conduct of research studies at MCI. This guidance will ensure the integrity of clinical data, compliance with the protocol and regulatory guidelines. This study will be monitored by University of South Alabama Mitchell Cancer Institute PI.

Study Title: Effects of a seven-day BASIS™ supplementation on menopausal syndromes and measurements of the urinary vitamin B3 and estradiol levels in pre-, peri- and post-menopause.

Risk Classification of the study:

For this study, there is intervention, and it is a minimal risk study.

The objectives of the monitoring are to:

1. Ensure subjects are being consented appropriately and prior to any study-related procedures.
2. Verify subject eligibility.
3. Ensure all adverse events are reported in a timely manner.
4. Audit data against source documents.
5. Verify maintenance of regulatory documents.
6. Verify study drug accountability.

Type of Research Data or Events to be Monitored:

The study data manager and the coordinating PI will keep up-to-date data on a regular basis. Accrual and safety data on this protocol will be reviewed by the PI, Data Manager, and Study Coordinator. Meetings will be held monthly for 3 months then held quarterly thereafter until completion of the study and End of Study meeting. The minutes of each meeting will be provided for review by IRB at the University of South Alabama for their independent review. All reports will be provided to the IRB of record and the study sponsor, Elysium Health.

Person(s) Responsible for Data Monitoring:

The purpose of monitoring is to ensure the rights of the human participants are protected, the clinical trial is conducted in compliance with established guidelines and protocol as well as to confirm that the data collected is accurate. Monitoring is performed by Dr. Marie Migaud, that is assigned to the study and familiar with the Protocol, Informed Consent, SOPs, etc.

Reporting Unanticipated Problems, Adverse Events, Protocol Deviations and Protocol Violations:

Protocol deviations are to be documented by the PI (Dr Migaud) using the Protocol Deviation Form and sent via e-mail to the IRB for review. Deviations that are considered major because they impact subject safety or alter the risk/benefit ratio, compromise the integrity of the study data, and/or affect subjects' willingness to participate in the study must be reported within 10 calendar days of awareness of the event.

The PI will be responsible for reporting adverse events experienced by participants under their care, untoward events occurring during the course of the study, protocol deviations and protocol violation by completing Protocol Deviation Forms and acknowledgments for regulatory filing to the sponsor. Protocol Deviations will be reported in monitoring reports:

* When the site is requesting a waiver or when a deviation from the protocol has occurred using the process noted above.
* The Sponsor Team (Elysium Health) and the IRB, in turn, review and respond to the deviation. At times, the Sponsor Team may request additional information from the site to clarify the deviation or waiver request.

Procedures and Time Frames for Communicating Outcomes:

Monitoring of the primary objective will be performed and reviewed for impact. Additionally, review of adverse events will occur monthly for the first 3 months and then quarterly thereafter until completion of the study. Possible Adverse Events will be reviewed by the Study's Clinical Principal and co-Principal Investigator

Emergency Actions:

Unblinding- This is not a blinded study.

Stopping Rules- This is a basic research study with no predefined endpoints other than data acquisition to support or invalidate a hypothesis.

The pre-defined safety-efficacy stopping points for the entire study that would cause the study to be suspended or terminated would be if there are concerns about the safety of the participant or about data integrity.

ELIGIBILITY:
Inclusion Criteria:

* 35 years of age or older
* pre, peri or post menopausal

Exclusion Criteria:

* Less than 35 years of age
* Hormone replacement therapy

Min Age: 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Biological female as determined at birth
Enrollment: 40 (Actual)
Dates: Start 2021-04-05 (Actual); Primary Completion 2021-07-15 (Actual); Study Completion 2021-07-15 (Actual)

PRIMARY OUTCOMES:
Production of Estradiol | 7 days
  To determine whether a short supplementation with BASIS™ impacts the natural production of estradiol, measured in urinary waste.
Change undesirable effects of menopause | 7 days
  To determine whether, through increased estradiol levels, the undesirable menopausal effects are impacted by a short-term supplementation with BASIS™.

CONTACTS AND LOCATIONS:
Locations (1):
- University of South Alabama, Mobile, Alabama, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Parazzini F. Resveratrol, tryptophanum, glycine and vitamin E: a nutraceutical approach to sleep disturbance and irritability in peri- and post-menopause. Minerva Ginecol. 2015 Feb;67(1):1-5. PMID 25660429
- [Result] Uberti F, Morsanuto V, Aprile S, Ghirlanda S, Stoppa I, Cochis A, Grosa G, Rimondini L, Molinari C. Biological effects of combined resveratrol and vitamin D3 on ovarian tissue. J Ovarian Res. 2017 Sep 15;10(1):61. doi: 10.1186/s13048-017-0357-9. PMID 28915830
- [Result] Davinelli S, Scapagnini G, Marzatico F, Nobile V, Ferrara N, Corbi G. Influence of equol and resveratrol supplementation on health-related quality of life in menopausal women: A randomized, placebo-controlled study. Maturitas. 2017 Feb;96:77-83. doi: 10.1016/j.maturitas.2016.11.016. Epub 2016 Nov 27. PMID 28041599
- [Result] Leo L, Surico D, Deambrogio F, Scatuzzi A, Marzullo P, Tinelli R, Molinari C, Surico N. [Preliminary data on the effectiveness of resveratrol in a new formulation in treatment of hot flushes]. Minerva Ginecol. 2015 Oct;67(5):475-83. Italian. PMID 26491826
- [Result] Narumi M, Takahashi K, Yamatani H, Seino M, Yamanouchi K, Ohta T, Takahashi T, Kurachi H, Nagase S. Oxidative Stress in the Visceral Fat Is Elevated in Postmenopausal Women with Gynecologic Cancer. J Womens Health (Larchmt). 2018 Jan;27(1):99-106. doi: 10.1089/jwh.2016.6301. Epub 2017 Aug 17. PMID 28816586
- [Result] Murugesan K, Vij U, Lal B, Farooq A. Effect of progestins, estradiol, and coenzymes NAD and NADPH on the interconversion of estradiol and estrone in rabbit uterus in vitro. Steroids. 1989 Jun;53(6):695-712. doi: 10.1016/0039-128x(89)90061-5. PMID 2554542
- [Result] Yaku K, Okabe K, Nakagawa T. NAD metabolism: Implications in aging and longevity. Ageing Res Rev. 2018 Nov;47:1-17. doi: 10.1016/j.arr.2018.05.006. Epub 2018 Jun 5. PMID 29883761
- [Result] Bonkowski MS, Sinclair DA. Slowing ageing by design: the rise of NAD+ and sirtuin-activating compounds. Nat Rev Mol Cell Biol. 2016 Nov;17(11):679-690. doi: 10.1038/nrm.2016.93. Epub 2016 Aug 24. PMID 27552971
- [Result] Joffe H, Petrillo LF, Koukopoulos A, Viguera AC, Hirschberg A, Nonacs R, Somley B, Pasciullo E, White DP, Hall JE, Cohen LS. Increased estradiol and improved sleep, but not hot flashes, predict enhanced mood during the menopausal transition. J Clin Endocrinol Metab. 2011 Jul;96(7):E1044-54. doi: 10.1210/jc.2010-2503. Epub 2011 Apr 27. PMID 21525161